CLINICAL TRIAL: NCT06502860
Title: Skin-to-Skin Contact With a Sling in Primipar Mothers Who Delivered by Cesarean Section
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Acibadem University (Other)
Responsible Party: Principal Investigator, Merve Coskun, Assistant Professor, Acibadem University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2024-5/171
Record Dates: First submitted 2024-07-09; First posted 2024-07-16 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Breast Feeding; Caesarean Section;Stillbirth
Keywords: Skin-to-skin contact; Caesarean section; Breastfeeding success; Newborn physiological weight loss; Sling
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Experimental Design
Who Masked: Participant
Masking Description: In the single-blind method, subjects do not know which of the experimental or control groups they were selected and therefore which method was applied to them. The researcher knows the subjects selected for the experimental and control groups, and therefore which method was applied to which subjects.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): The intervention group will receive skin-to-skin contact facilitated by the use of a sling. Immediately after the cesarean section and stabilization, the newborn will be placed against the mother's bare chest using a specially designed sling. This sling will secure the baby in a safe and comfortable position, allowing for continuous close contact. The duration of skin-to-skin contact will be encouraged to last as long as the mother and baby are comfortable, without any set time limits.
  Interventions: Other: skin to skin with sling
- Control Group (No Intervention): The control group will receive standard skin-to-skin contact without the use of a sling. Immediately after the cesarean section and stabilization, the newborn will be placed directly on the mother's bare chest. This traditional method will involve holding the baby manually to maintain skin-to-skin contact. The duration of skin-to-skin contact will be encouraged to last as long as the mother and baby are comfortable, without any set time limits.

INTERVENTIONS:
Other: skin to skin with sling — In the intervention group, skin-to-skin contact will be facilitated using a specially designed sling. This approach aims to enhance the quality and duration of skin-to-skin contact between the mother and the newborn.
  Arms: Experimental Group

SUMMARY:
The first hours after birth are critical for the physiological and psychological adaptation process of the newborn from intrauterine to extrauterine life. The World Health Organization (WHO) recommends skin-to-skin contact as a routine part of care to stabilize the newborn's vital signs and strengthen the mother-infant bond. However, the rate of skin-to-skin contact in women who give birth by cesarean section is lower compared to vaginal deliveries. Considering the global increase in cesarean birth rates, it is necessary to develop appropriate and practical care methods for mothers and newborns who deliver by cesarean section.

The literature has examined the effects of the duration of skin-to-skin contact on breastfeeding initiation, neonatal hypothermia, and cardiopulmonary stability. However, studies aimed at increasing the duration of skin-to-skin contact are limited. This study compares the effects of standard skin-to-skin contact and skin-to-skin contact using a sling on the duration of skin-to-skin contact, postpartum breastfeeding success, and physiological weight loss of the newborn in primiparous mothers who delivered by cesarean section.

ELIGIBILITY:
Inclusion Criteria:

* Healthy mothers who gave birth by cesarean section
* Primiparous mothers
* Healthy newborns

Exclusion Criteria:

* Mothers who gave birth vaginally
* Newborns using formula milk
* Mothers with breastfeeding difficulties
* Preterm newborns
* Multiple births
* Mothers and newborns with unstable health conditions

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2024-09-15 (Actual); Primary Completion 2025-08-11 (Actual); Study Completion 2025-08-11 (Actual)

PRIMARY OUTCOMES:
Introductory Information Form | Baseline (to both groups before the intervention)
  The introductory characteristics of the mother and newborn are documented in forms used by the institution during patient care and in records. These forms are created by the researchers to systematize the information used in this study.
Skin-to-Skin Contact Tracking Form | To be completed during patient follow-up (postpartum days 0, 1, and 2)
  This form is created by the researchers to determine the duration of skin-to-skin contact for each participant.
Breastfeeding Assessment Scale (LATCH) | To be completed during patient follow-up, once a day (postpartum days 0, 1, and 2)
  The scale, developed by Jensen and Wallace in 1993, aims to objectively assess breastfeeding, identify breastfeeding problems, plan education, establish a common language among healthcare professionals, and be used in research (Jensen et al., 1994). The scale was adapted into Turkish by Yenal and Okumuş in 2003 and consists of five assessment steps. It is modeled after the APGAR scoring system and is quick and easy to use. The acronym LATCH stands for the English terms of these assessment steps: "L = Latch on breast," "A = Audible swallowing," "T = Type of nipple," "C = Comfort breast/nipple," "H = Hold." Each item is scored between 0-2 points. The total possible score from the measurement tool is 10. There is no cut-off point for the tool. As the LATCH score increases, the success of breastfeeding is understood to be higher. The scale has a Cronbach alpha value of .95 (Yenal and Okumuş, 2003).

CONTACTS AND LOCATIONS:
Locations (1):
- Merve Coşkun, Ataşehir, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF, CSR
Time Frame: after the publication
Access Criteria: Online database link will be sent

REFERENCES:
- [Result] Takahashi Y, Tamakoshi K, Matsushima M, Kawabe T. Comparison of salivary cortisol, heart rate, and oxygen saturation between early skin-to-skin contact with different initiation and duration times in healthy, full-term infants. Early Hum Dev. 2011 Mar;87(3):151-7. doi: 10.1016/j.earlhumdev.2010.11.012. Epub 2011 Jan 8. PMID 21220191
- [Result] Wigglesworth H, Huddy V, Knowles R, Millings A. Evaluating the impact of sling provision and training upon maternal mental health, wellbeing and parenting: A randomised feasibility trial. PLoS One. 2023 Nov 10;18(11):e0293501. doi: 10.1371/journal.pone.0293501. eCollection 2023. PMID 37948400
- [Result] Kollmann M, Aldrian L, Scheuchenegger A, Mautner E, Herzog SA, Urlesberger B, Raggam RB, Lang U, Obermayer-Pietsch B, Klaritsch P. Early skin-to-skin contact after cesarean section: A randomized clinical pilot study. PLoS One. 2017 Feb 23;12(2):e0168783. doi: 10.1371/journal.pone.0168783. eCollection 2017. PMID 28231274
- [Result] Gouchon S, Gregori D, Picotto A, Patrucco G, Nangeroni M, Di Giulio P. Skin-to-skin contact after cesarean delivery: an experimental study. Nurs Res. 2010 Mar-Apr;59(2):78-84. doi: 10.1097/NNR.0b013e3181d1a8bc. PMID 20179657